CLINICAL TRIAL: NCT05311540
Title: Zinc Supplementation In Very Low Birth Weight Infants-A Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Suzan Sahin, Specialist, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: ZincVLBW
Record Dates: First submitted 2019-05-19; First posted 2022-04-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Preterm Infant; Effect of Drugs; Zinc Deficiency Disease
MeSH Terms: conditions — Premature Birth | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An independent physician not involved in the study conducted the random assignment process. The investigators who were blinded to the randomisation process closely followed up the enrolled infants for any evidence of feeding intolerance and/or NEC, late-onset sepsis (LOS), bronchopulmonary dysplasia (BPD), hemodynamically significant patent ductus arteriosus (hsPDA), intraventricular hemorrhage (IVH), retinopathy of prematurity (ROP) along with other possible neonatal morbidities and signs of toxicity or side effects (adverse events)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc intervention (Experimental): 9 mg/day Zinc suspension via og tube along with the routinely used standard multivitamin product containing 3 mg daily dose of Zn, started on day 7 until discharge from hospital
  Interventions: Drug: Zinc Sulfate
- Control (No Intervention): These infants received only standard commercial multivitamin product containing 3 mg daily dose of Zn

INTERVENTIONS:
Drug: Zinc Sulfate
  Arms: Zinc intervention

SUMMARY:
* Zinc (Zn) is a structural component of human body and is a crucial element for a wide variety of cascades that take place in almost all organ systems.
* Due to many reasons, preterm infants are generally believed to be naturally in a negative Zn balance during the early periods of life.
* Regulation of intestinal Zn absorption of preterms is unrelated to infant's Zn status.
* There still is a lack of knowledge in the possible relation of Zn deficiency and development of NEC and/or feeding intolerance in preterm infants.
* Even if Zn is studied as an adjunct treatment for neonates and young infants with sepsis and found to reduce treatment failure in these high risk population, data in preventing infectious diseases in preterm infants is still lacking.

DETAILED DESCRIPTION:
Background and Objectives: Preterm infants have high zinc (Zn) requirements and are generally believed to be in a negative Zn balance in the early period of life. In this study, we aimed to investigate the effect of high dose Zn supplementation in very low birth weight (VLBW) infants on feeding intolerance and development of mortality and/or morbidities including necrotizing enterocolitis (NEC), late-onset sepsis (LOS).

Methods: This is a prospective randomized trial. VLBW preterm infants with gestational age of <32 weeks were randomly allocated on the seventh day of life to receive extra amount of supplemental zinc along with the enteral feedings or not, besides regular low dose supplementation, from enrollment until discharge. Outcome measures were feeding intolerance, NEC (stage≥2), LOS and mortality.

ELIGIBILITY:
Inclusion Criteria:

* < 32 weeks gestational age and/or <1500 gr birth weight
* Born in the study hospital
* Being able to be fed enterally, even in very small amounts, regardless of the volume of the nutrient

Exclusion Criteria:

* Major congenital malformations and/or critical congenital heart defects
* Born in another hospital
* Severe birth asphyxia
* Severe sepsis
* Previous early-onset NEC history
* Infants on the intervention arm who did not continue Zinc supplementation during the study period
* Hemodynamically unstability
* Infants nil per os
* No consent from the family
* Death before the 7th day of life

Ages: 7 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2015-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of feeding intolerance | through study completion, an average of 6 months

SECONDARY OUTCOMES:
Duration of hospitalization | through study completion, an average of 6 months
Number of participants with necrotising enterocolitis (stage≥2) | through study completion, an average of 6 months
Incidence of mortality | through study completion, an average of 6 months
Number of participants with late onset sepsis | through study completion, an average of 6 months
Number of participants with retinopathy of prematurity | through study completion, an average of 6 months
Number of participants with bronchopulmonary dysplasia | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Democracy University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No